CLINICAL TRIAL: NCT05110495
Title: Windows Trial of INsulin-like Growth Factor Neutralising Antibody Xentuzumab in MEN Scheduled for Radical Prostatectomy (WINGMEN)
Brief Title: IGF Inhibition With Xentuzumab Prior to Radical Prostatectomy
Acronym: WINGMEN
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Prostate Cancer UK (Other); Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OCTO-084
Record Dates: First submitted 2021-08-23; First posted 2021-11-08 (Actual); Results first posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2024-07

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — xentuzumab

STUDY DESIGN:
Intervention Model Description: This is a phase 0 'window of opportunity' study testing whether xentuzumab blocks IGF signalling and markers of growth in men with localised prostate cancer scheduled for radical prostatectomy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Xentuzumab (Experimental): All patients will be allocated to receive Xentuzumab
  Interventions: Drug: Xentuzumab

INTERVENTIONS:
Drug: Xentuzumab — The study IMP is xentuzumab, a humanised IgG1 monoclonal antibody that neutralises the IGF ligands to inhibit activation of IGF-1R and INSR-A, suppressing IGF-mediated proliferation, invasion and therapy resistance

SUMMARY:
The WINGMEN trial aims to understand how a hormone-like protein called insulin-like growth factor (IGF) helps prostate cancers grow and become aggressive. IGF is required for normal development, and also helps cancers grow and spread. Men with high blood IGF are at increased risk of developing prostate cancer, and tall men are more likely to get aggressive prostate cancer. The WINGMEN trial will recruit 30 men with prostate cancer who have been offered an operation to remove the prostate. Most men have to wait 4-5 weeks between a decision to have prostate removal surgery, and actually having the operation. In this 4-5 week window we will offer treatment with a new IGF-blocker drug called xentuzumab. The drug is provided by Boehringer Ingelheim and the trial is funded by Prostate Cancer UK.

Xentuzumab will be given as an outpatient by once weekly intravenous infusion (drip) in the Early Phase Clinical Trials Unit, Oxford Cancer Centre, Churchill Hospital. In other trials, xentuzumab is being tested in patients with advanced cancer, and is proving to be well-tolerated. After the 4-week treatment, WINGMEN trial patients will have routine prostate removal surgery. Samples of blood and prostate cancer that are surplus to diagnostic need will be taken from the diagnostic prostate biopsy (pre-xentuzumab) and the cancer removed at surgery (after xentuzumab) for research tests. These samples will be compared to measure how effectively xentuzumab reduces signs of tumour growth, and identify which genes and proteins are switched on or off by xentuzumab, and which may therefore be important in helping IGF promote prostate cancer growth. The information we get from the WINGMEN trial may help us to improve treatment of men with prostate cancer, with the long-term aim of reducing the risk of aggressive prostate cancer

ELIGIBILITY:
Inclusion Criteria:

A patient will be eligible for inclusion in this study if all of the following criteria apply.

1. Men with prostate adenocarcinoma confirmed on prostate biopsy and with sufficient cancer-containing biopsy tissue surplus to diagnostic need to provide 2 sections for primary endpoint analysis.
2. Scheduled for open or robotic radical prostatectomy
3. Age ≥ 18 years
4. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1 (Appendix 1)
5. The patient is willing and able to comply with the protocol scheduled follow-up visits and examinations for the duration of the study
6. Participant is willing and able to give informed consent.
7. Participants whose partner is of child bearing potential must be willing to ensure that they or their partner use effective contraception during the trial and for 70 days thereafter.
8. Adequate hematologic, renal and hepatic function, defined as follows:

Laboratory Test Value required Hemoglobin (Hb) ≥90g/L White Blood Count (WBC) >2.5 x 10*9/L Absolute Neutrophil Count (ANC) ≥ 1.5 x10*9/L Platelet count ≥ 100 x 10*9/L AST, ALT, and alkaline phosphatase ≤ 2.5 x upper limit of normal eGFR* ≥30ml/min

*eGFR calculated by Cockcroft & Gault formula,

Exclusion Criteria:

* A patient will not be eligible for the trial if any of the following apply:

  1. Treated with systemic corticosteroids, insulin, metformin, other oral hypoglycemic agent, or anti-androgens in the 28 days prior to first dose of study drug
  2. Diabetes mellitus
  3. Previous prostate radiotherapy
  4. Current or previous treatment with xentuzumab or other IGF or GH -modifying therapy
  5. Patients who are known to be serologically positive for Hepatitis B, Hepatitis C or HIV
  6. Treatment with any other investigational agent, or treatment in another interventional clinical trial within 28 days prior to enrolment
  7. Other psychological, social or medical condition, physical examination finding or a laboratory abnormality that the Investigator considers would make the patient a poor trial candidate or could interfere with protocol compliance or the interpretation of trial results

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — based on gender identity
Enrollment: 27 (Actual)
Dates: Start 2021-12-17 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simon Lord, Prof, Principal Investigator — University of Oxford
Locations (1):
- Churchill Hospital, Oxford University Hospitals, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Xentuzumab
Started | 27
Completed | 25
Not Completed | 2
Not completed — Lost to Follow-up | 1
Not completed — Completed treatment with IMP but disease progressed prior to surgery. | 1

BASELINE CHARACTERISTICS:
Arm/Group | Xentuzumab
Number analyzed (Participants) | 27
Age, Continuous [Median (Full Range); unit: years] | 66 [50 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 27

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change of Phospho-IGF-1R Positive Tumour Cells Following Treatment With Xentuzumab
Description: Diagnostic biopsies (pre-treatment) and in-theatre cores (post-treatment) were stained with phospho-IGF-1R. Percentage of positively stained tumour cells in each sample were compared and the percentage change between timepoints was quantified. A negative percentage change indicates a reduction in phospho-IGF-1R in post-treatment samples. This endpoint was designed to assess the amount of IGF pathway inhibition induced by xentuzumab.
Time Frame: From first xentuzumab infusion at week 1 (pre-treatment) to surgery at week 4-13 (post-treatment). Up to 13 weeks total.
Population: Units given accounts for a pre-treatment and post-treatment sample per participant. Number analysed excludes samples from 6 participants that were missing either the pre-treatment or post-treatment sample, or could not be analysed for other reasons.
Measure: Mean (Full Range); unit: Percentage change Phospho-IGF-1R+ cells
Units Other Than Participants: Tissue samples
Arm/Group | Xentuzumab
Number analyzed (Participants) | 21
Number analyzed (Tissue samples) | 42
Percentage change Phospho-IGF-1R+ cells | -8.28 [-97.94 to 481.68]

2. Primary Outcome: Percentage Change of Phospho-S6 Positive Tumour Cells Following Treatment With Xentuzumab
Description: Diagnostic biopsies (pre-treatment) and in-theatre cores (post-treatment) were stained by phospho-S6. Percentage of positively stained tumour cells in each sample were compared and the percentage change between timepoints was quantified. A negative percentage change indicates a reduction in phospho-S6 in post-treatment samples. This endpoint was designed to assess the amount of IGF pathway inhibition induced by xentuzumab.
Time Frame: From first xentuzumab infusion at week 1 (pre-treatment) to surgery at week 4-13 (post-treatment). Up to 13 weeks total.
Population: Units analysed describes pre-treatment and post-treatment sample for each participant. Number analysed excludes 10 participants that were missing either the pre-treatment or post-treatment sample, or could not be analysed for other reasons.
Measure: Mean (Full Range); unit: Percentage change of Phospho-S6+ cells
Units Other Than Participants: Tissue samples
Arm/Group | Xentuzumab
Number analyzed (Participants) | 17
Number analyzed (Tissue samples) | 34
Percentage change of Phospho-S6+ cells | -52.55 [-87.61 to 60.11]

3. Secondary Outcome: Number of Participants Who Had at Least 4 Doses of Xentuzumab and Proceeded to Have Surgery Per the Protocol Schedule
Description: This endpoint was a measure of feasibility of the treatment schedule in the pre-operative setting.
Time Frame: From first xentuzumab infusion at week 1 (pre-treatment) to surgery at week 4-13 (post-treatment). Up to 13 weeks total.
Population: Total number of participants who had at least 4 doses of xentuzumab. Excludes one registered patient who progressed prior to surgery and came off trial.
Measure: Count of Participants; unit: Participants
Arm/Group | Xentuzumab
Number analyzed (Participants) | 26
Participants
  Surgery performed on schedule | 26
  Surgery delayed by trial treatment | 0

4. Secondary Outcome: Median Delay in Surgery in Participants Who Had More Than 4 Doses of Xentuzumab (and Whose Surgery Was Delayed by Factors Other Than Trial Treatment)
Description: All participants who had more than 4 doses of xentuzumab were considered to have had their surgery delayed by factors other than trial treatment. Per protocol, all participants who had delayed surgery received additional weekly doses of xentuzumab. Reason for delay was not recorded as part of the study dataset. This endpoint was a measure of feasibility of the treatment schedule in the pre-operative setting.
Time Frame: From first xentuzumab infusion at week 1 (pre-treatment) to surgery at week 4-13 (post-treatment). Up to 13 weeks total.
Population: Number of participants who had more than 4 Doses of xentuzumab.
Measure: Median (Full Range); unit: weeks
Arm/Group | Xentuzumab
Number analyzed (Participants) | 15
weeks | 2 [2 to 9]

5. Secondary Outcome: Number of Patients Experiencing an Adverse Event (AE) or Serious Adverse Event (SAE) While On-trial
Description: This endpoint was designed to assess safety and tolerability of xentuzumab administered in the pre-prostatectomy setting. AEs & SAEs were graded using CTCAE v5.0, with higher grades considered to be worse outcomes.
Time Frame: From consent at week -1 to the end of study visit at up to 19 weeks
Population: All participants registered to take part in the WINGMEN trial. All participants received xentuzumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Xentuzumab
Number analyzed (Participants) | 27
Participants
  Any AE, Highest Grade 1 or 2 (CTCAE v5.0) | 23
  Any AE, Highest Grade 3,4,5 (CTCAE v5.0) | 1
  Any SAE, Highest Grade 1 or 2 (CTCAE v5.0) | 0
  Any SAE, Highest Grade 3,4,5 (CTCAE v5.0) | 0
  No AEs or SAEs reported | 3

6. Secondary Outcome: Number of Patients With Any Adverse Event Assessed as Treatment-Related (TRAE) While On-trial
Description: Number of patients with any TRAE from the time of consent to the end of study visit. TRAEs are AEs that are investigator-determined to be definitely, probably or possibly related to treatment with xentuzumab and graded using CTCAE v5.0, with higher grades considered to be worse outcomes.
  This endpoint was designed to assess safety and tolerability of xentuzumab administered in the pre-prostatectomy setting.
Time Frame: From consent at week -1 to the end of study visit at up to 19 weeks
Population: All participants registered to take part in the WINGMEN trial. All participants received xentuzumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Xentuzumab
Number analyzed (Participants) | 27
Participants
  Any TRAE, Highest Grade 1 or 2 (CTCAE v5.0) | 17
  Any TRAE, Highest Grade 3,4,5 (CTCAE v5.0) | 0
  No TRAE | 10

ADVERSE EVENTS:
Time Frame: From consent to end of study visit (up to 19 weeks).
Description: Adverse Event data was collected during trial visits from investigator-led assessments as specified in the protocol.
Groups:
- Xentuzumab: All patients were allocated to receive the study IMP, Xentuzumab. Xentuzumab is a humanised IgG1 monoclonal antibody that neutralises the IGF ligands to inhibit activation of IGF-1R and INSR-A, suppressing IGF-mediated proliferation, invasion and therapy resistance.
Arm/Group | Xentuzumab
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 24/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Xentuzumab (N=27)
Blood & Lymphatic System Disorders (Blood and lymphatic system disorders) | 5 (10)
Eye disorders (Eye disorders) | 1 (1)
Gastrointestinal Disorders (Gastrointestinal disorders) | 8 (12)
General Disorders & Administration Site Conditions (General disorders) | 11 (15)
Infections & Infestations (Infections and infestations) | 5 (6)
Injury; poisoning and procedural complications (Injury, poisoning and procedural complications) | 3 (3)
Metabolism & Nutrition Disorders (Metabolism and nutrition disorders) | 4 (5)
Musculoskeletal & Connective Tissue Disorders (Musculoskeletal and connective tissue disorders) | 7 (7)
Nervous System Disorders (Nervous system disorders) | 6 (8)
Renal and urinary disorders (Renal and urinary disorders) | 11 (13)
Reproductive system and breast disorders (Reproductive system and breast disorders) | 3 (3)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 2 (2)
Surgical and medical procedures (Surgical and medical procedures) | 3 (3)
Vascular disorders (Vascular disorders) | 3 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-11-21): https://cdn.clinicaltrials.gov/large-docs/95/NCT05110495/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-24): https://cdn.clinicaltrials.gov/large-docs/95/NCT05110495/SAP_001.pdf